CLINICAL TRIAL: NCT02507531
Title: INCA: Intracranial Aneurysm Treatment With NeXsys
Acronym: INCA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Cerus Endovascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNX-041
Record Dates: First submitted 2015-07-20; First posted 2015-07-24 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2016-05

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Placement of study device (currently called NeXsys) into target aneurysm via standard endovascular procedure.
  Interventions: Device: NeXsys Embolization System

INTERVENTIONS:
Device: NeXsys Embolization System — Woven metallic mesh placed in aneurysm fundus
  Other Names: Contour Neurovascular System

SUMMARY:
Prospective, single center first-in-man study of use of device for intracranial aneurysm occlusion

DETAILED DESCRIPTION:
Prospective, single center first-in-man study of use of device for intracranial aneurysm occlusion. Target aneurysms are small unruptured aneurysms in the anterior and posterior circulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years at screening
* Unruptured saccular IA in the anterior or posterior circulation with dimensions consistent with Table 2
* IA appears suitable for NeXsys device
* Patient willing to comply with study requirements
* Patient able to understand and sign a study-specific informed consent form

Exclusion Criteria:

* Ruptured IA
* Any other IA that requires treatment in the next year
* IA width >10 mm
* IA neck >9 mm
* IA has important flow from its base such that occluding the IA would cause stroke
* Target IA contains any device (e.g., coils)
* Inability to access the target IA with microcatheter
* Any congenital or iatrogenic coagulopathy
* Platelet count <50,000/microliter
* Known allergy to platinum, nickel or titanium
* Known allergy to contrast agents
* Stenosis of the target IA's parent vessel >50%
* Taking daily aspirin or other platelet inhibitor (clopidogrel or equivalent)
* Taking any anticoagulants (e.g., warfarin)
* Pregnant or planning pregnancy in the next 2 years
* Other medical conditions that could increase the risk of neurovascular procedures (e.g., liver failure, cancer, etc.)
* Participating in another study with investigational devices or drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-05; Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Safety: occurrence of major ipsilateral stroke or neurologic death | 3-6 months
Ability of the investigator to place the device in an acceptable position in the target IA, judged at the time of placement, with no migration or change in position of the device at 3-6 month angiogram. | 3-6 mo

SECONDARY OUTCOMES:
Occlusion status of the target IA at 30 days, 3-6 months, 1 year and 5 years as judged by an independent physician using the Raymond classification system. | 30 days, 3-6 months, 1 year and 5 years
Occurrence rate of any neurologic or vascular adverse event related to the target IA or device placement procedure | Beginning of index procedure to end of index procedure (approximately 1 hour, maximum 3 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Clinico ENERI, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided